CLINICAL TRIAL: NCT06429306
Title: A Phase 3,Prospective, Randomized, Double-masked, Placebo-controlled, Parallel Study to Evaluate the Efficacy, PK and Safety of 9% Dexamethasone Intraocular Injection for the Treatment of Inflammation Associatedwith Cataract Surgery
Brief Title: Study of Dexycu in Treating Intraocular Inflammation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ocumension Therapeutics (Shanghai) Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Ocumension Therapeutics (Suzhou) Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OT-502-001
Record Dates: First submitted 2024-05-11; First posted 2024-05-24 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Inflammation; Cataract
Keywords: Cataract Surgery; Postoperative Inflammation
MeSH Terms: conditions — Inflammation; Cataract | interventions — Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dexamethasone intraocular injection (Experimental): Dexamethasone implant single injection in the treatment eye after cataract surgery.
  Interventions: Drug: Dexycu
- Placebo (Placebo Comparator): Blank placebo single injection in the treatment eye after cataract surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexycu — 5ul dexamethasone, concentration: 103.4 μg/μl, equivalent to 517μg dexamethasone
  Other Names: Investigational product
  Arms: Dexamethasone intraocular injection
Drug: Placebo — Acetyl triethyl citrate
  Arms: Placebo

SUMMARY:
This is a phase III, prospective, randomised, double-masked, placebo-controlled, parallel-design, multicenter study of the efficacy, safety and pharmacokinetics of 9% dexamethasone intraocular injection for the treatment of inflammation associated with cataract surgery.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blindmasked, placebo-controlled, parallel- design, multicenter study of subjects over 40 years undergoing cataract surgery. Subjects meet the inclusion criteria and do not meet any exclusion criteria are randomiszed to the dexamethasone implant group or placebo group at a ratio of 2:1.

Subjects received a single does injection in the study eye immediately after the completion of cataract surgery. The investigational drug comes with a special injection device and injection guide.

All subjects will be administered to the study eye with quinolone topical antibiotic eye drops or their equivalent 3 days before and 7 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must provide written informed consent by signing the Informed Consent approved by the Institutional Review Board (IRB).
2. Male or female patients at least 40 years of age scheduled for unilateral cataract surgery by phacoemulsification with posterior chamber intraocular lens implantation.
3. The patient must demonstrate best corrected visual acuity (BCVA) of 20/30-20/200 in the study eye and better than 20/200 in the fellow eye.
4. The patient must be considered by the Investigator to have visual acuity potential. greater than 20/30 in the study eye.
5. The patient must have a corneal endothelial cell count by specular microscopy in the study eye of at least 2000 cells/mm2 with normal cell morphology.
6. A female patient of childbearing potential must have a negative pregnancy test on Day 0 and be using an effective method of birth control from Screening for the duration of the study.
7. The patient must be willing and able to understand and comply with the study procedures and to communicate meaningfully with study personnel.

Exclusion Criteria:

1. Patients who have used any ocular, topical or oral corticosteroids within 7 days prior to Day 0.
2. Patients who have received a periocular corticosteroid injection in the study eye in the 3 months prior to screening.
3. Patients who have received any intravitreal corticosteroid delivery vehicle (e.g.,Retisert, Ozurdex, Iluvien) in the study eye at any time.
4. Patients who anticipate requiring treatment with any corticosteroids( by any route,except inhalation), during the study.
5. Patients with an allergy or hypersensitivity to dexamethasone.
6. Patients who are known steroid responders (corticosteroid-related intraocular pressure elevation in either eye).
7. Patients who have used topical ocular NSAIDs in the study eye within 15 days prior to Day 0.
8. Patients who have undergone prior intraocular (non-laser) surgery in the study eye within 6 months prior to screening.
9. Patients who have undergone prior intraocular laser surgery in the study eye within 3 months prior to screening.
10. Patients with planned intraocular or laser surgery in the study eye for the duration of the study.
11. Patients with any signs of intraocular inflammation in either eye at screening.
12. Patients with evidence of corneal abnormality or dystrophy (e.g. opacities, guttae,clouding, etc.) or an inability to obtain an acceptable specular micrograph at Screening.
13. Patients with a history of chronic uveitis from any cause in either eye.
14. Patients who have received any prior intravitreal injections in the study eye.
15. Patients with glaucomatous optic neuropathy or glaucomatous visual field loss in either eye.
16. Patients with ocular hypertension with an IOP in the study eye > 21 mm Hg at Screening with or without treatment with anti-glaucoma monotherapy.
17. Patients with ocular hypertension receiving treatment with two or more anti-glaucoma Medications.
18. Patients treated with any investigational product within 30 days prior to screening or patients enrolled previouslyc study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2022-08-22 (Actual); Primary Completion 2023-11-24 (Actual); Study Completion 2024-04-09 (Actual)

PRIMARY OUTCOMES:
Anterior chamber cell clearing rate | DAY 8
  The primary efficacy outcome is anterior chamber cell clearing in the study eye at Day 8. The slit lamp examination for anterior chamber cells (ACC) is a recognized way to measure inflammation in the anterior chamber. During the slit lamp examination, the number of anterior chamber cells are quantified and graded: grade 0 (absent, 0 cells), grade 1 (1 to 5 cells), grade 2 (6 to 15 cells), grade 3 (16 to 30+ cells), or grade 4 (hypopyon). Anterior chamber cell clearing occurs when all the ACC are absent (grade 0).

SECONDARY OUTCOMES:
Anterior chamber cell clearing rates | DAY 1 & 3 & 15 & 30
  The secondary efficacy outcome is anterior chamber cell clearing in the study eye at Day 1 & 3 & 15 & 30. The slit lamp examination for anterior chamber cells (ACC) is a recognized way to measure inflammation in the anterior chamber. During the slit lamp examination, the number of anterior chamber cells are quantified and graded: grade 0 (absent, 0 cells), grade 1 (1 to 5 cells), grade 2 (6 to 15 cells), grade 3 (16 to 30+ cells), or grade 4 (hypopyon). Anterior chamber cell clearing occurs when all the ACC are absent (grade 0).
Anterior chamber flare clearing rates | DAY 1 & 3 & 8 & 15 & 30
  Percentage of subjects with anterior chamber flare grade 0 at Day 1, 3, 8, 15, and 30. The slit lamp examination for anterior chamber flare (ACF) is a recognized way to measure inflammation in the anterior chamber. During the slit lamp examination, the number of anterior chamber cells are quantified and graded: grade 0 (absent), grade 1 (trace), grade 2 (mild intensity), grade 3 (moderate intensity), or grade 4 (strong intensity). Anterior chamber flare clearing occurs when all the ACC are absent (grade 0).
Anterior chamber cell & flare clearing rates | DAY 1 & 3 & 15 & 30
  The secondary efficacy outcome is anterior chamber cell & flare clearing in the study eye at Day 1 & 3 & 15 & 30. The slit lamp examination for anterior chamber cells & flare (ACCF) is a recognized way to measure inflammation in the anterior chamber.
Mean anterior chamber cell score and mean anterior chamber flare score | DAY 8 & 15
  Calculate the mean score of anterior chamber cell and flare separately at Day 8 and 15.
Mean anterior chamber cell + flare score | DAY 8 &15
  Calculate the mean socre of anterior chamber cell + flare at Day 8 and 15.

CONTACTS AND LOCATIONS:
Overall Officials: Zhixun Li, Study Director — Ocumension Therapeutics (Shanghai) Co., Ltd
Locations (1):
- Shanghai General Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No